CLINICAL TRIAL: NCT06151600
Title: A Prospective Natural History and Outcome Measure Discovery Study of Charcot-Marie-Tooth Disease, Type 4J
Acronym: CMT4J
Status: Recruiting | Type: Observational
Sponsor: Elpida Therapeutics SPC (Industry)
Responsible Party: Sponsor
Other Study IDs: ELPIDA THERAPEUTICS CMT4J NHS
Record Dates: First submitted 2023-10-23; First posted 2023-11-30 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Peripheral Neuropathy; Neuro-Degenerative Disease; Neuromuscular Diseases
MeSH Terms: conditions — Peripheral Nervous System Diseases; Neuromuscular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples and skin biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a multicenter, longitudinal, prospective observational natural history study of subjects with a molecularly confirmed diagnosis of CMT4J. The study will enroll 20 subjects of any age into a uniform protocol for follow-up and evaluations. Subject visits will occur every 12 months + 4 weeks for up to 2 years.

DETAILED DESCRIPTION:
This is a multicenter, longitudinal, prospective observational natural history study of subjects with a molecularly confirmed diagnosis of CMT4J. The study will enroll 20 subjects of any age into a uniform protocol for follow-up and evaluations. The study will obtain demographic and medical history information. Natural history data will be collected prospectively on an annual basis and may include physical/neurological exams, standard laboratory tests, CMT outcome and disability measures, neuropsychological tests, nerve conduction studies (NCS), and imaging studies (muscle MRI). Pulmonary function test (PFT) and scoliosis series x-ray Subject visits will occur every 12 months + 4 weeks for up to 2 years. Subjects who terminate from the study prior to Visit 3 will undergo an early termination/end of study visit (EOS) if possible. The early termination/end of study visit is comprised of the Visit 3 assessments. If needed, the Investigator may conduct unscheduled visits with Sponsor's approval. No investigational product will be used during the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, all ages
2. A molecularly-confirmed diagnosis of CMT4J (confirmed by a CLIA certified, CE-marked, or equivalent lab): Genomic DNA mutation analysis demonstrating 1) bi-allelic pathogenic and/or likely pathogenic variants (by ACMG criteria) in the FIG4 gene, or 2) bi-allelic variants with one pathogenic and/or likely pathogenic variant in trans with a variant of uncertain significance if laboratory evidence and expert consensus exits in support of loss of FIG4 function exists.
3. Informed consent from patients 18 years or older who are able to provide consent and from caregivers; parent(s)/guardian(s) providing consent for subjects younger than 18 years at Screening and patients older than 18 years unable to provide informed consent
4. Informed assent of patients younger than 18 years at Screening who are able to provide assent
5. Able and willing to comply with the study protocol, including travel to Study Center, procedures, measurements and visits

Exclusion Criteria:

1. Any known genetic abnormality, including chromosomal aberrations that confound the clinical phenotype
2. Current participation in an interventional or therapeutic study
3. Receiving an investigational drug within 90 days of the Baseline Visit
4. Prior or current treatment with gene or stem cell therapy
5. Any other diseases which may significantly interfere with the assessment of CMT4J
6. Have any other conditions, which, in the opinion of the Investigator or Sponsor would make the subject unsuitable for inclusion or could interfere with the subject participating in or completing the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with a genetically confirmed diagnosis of CMT4J will be included.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-07-29 (Actual); Primary Completion 2031-03-01 (Estimated); Study Completion 2032-03-01 (Estimated)

PRIMARY OUTCOMES:
Study objective | 2 years
  This study is designed to investigate the clinical characteristics and natural history of CMT4J.

CONTACTS AND LOCATIONS:
Overall Officials: Souad Messahel, Ph.D, Study Director — Elpida Therapeutics SPC
Locations (3):
- United States (3):
  - Stanford University, San Francisco, California
  - University of Iowa, Iowa City, Iowa
  - University of Texas Southwestern, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
De-identified data for publication.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Starting in January 2025
Access Criteria: All Investigators leading the trial.

DOCUMENTS (1):
  • Study Protocol (2023-08-01): https://cdn.clinicaltrials.gov/large-docs/00/NCT06151600/Prot_000.pdf